CLINICAL TRIAL: NCT04208594
Title: Efficacy of Ivabradine Versus Propranolol Premedication During Hypotensive Anesthesia in Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Mohamed Osman, assistant professor of anesthesia Alexandria university, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Ivabradine; Propranolol; Hypotensive Anesthesia
MeSH Terms: interventions — Ivabradine; Propranolol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP (P): (Active Comparator): will receive oral propranolol (INDERAL® -propranolol hydrochloride Ph. Eur. 10mg manufactured by AstraZeneca Egypt under license of AstraZeneca UK), 10 mg one tablet at 8:00 pm in the evening before the day of the surgery and one 10 mg tablet one hour before the induction of anesthesia.
  Interventions: Drug: Propranolol
- GROUP (I): (Experimental): will receive oral ivabradine (Procoralan® 5mg manufactured by Servier laboratories, France), 5 mg one tablet at 8:00 pm in the evening before the day of the surgery and one 5 mg tablet one hour before the induction of anesthesia.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — comparing between both drugs for the effect of hypotensive anesthesia
  Arms: GROUP (I):
Drug: Propranolol — comparing between both drugs for the effect of hypotensive anesthesia
  Arms: GROUP (P):

SUMMARY:
50 Patients, aged from 18 to 39 years, ASA physical status I and II, undergoing endoscopic sinus surgery will be enrolled in the study.The patients will be randomly allocated by simple randomization using a computer programme into two groups by closed envelope technique (having 25 patients in each group): GROUP (P): will receive oral propranolol (INDERAL® -propranolol hydrochloride Ph. Eur. 10mg manufactured by AstraZeneca Egypt under license of AstraZeneca UK), 10 mg one tablet at 8:00 pm in the evening before the day of the surgery and one 10 mg tablet one hour before the induction of anesthesia.

GROUP (I): will receive oral ivabradine (Procoralan® 5mg manufactured by Servier laboratories, France), 5 mg one tablet at 8:00 pm in the evening before the day of the surgery and one 5 mg tablet one hour before the induction of anesthesia.

DETAILED DESCRIPTION:
Aim of the work To compare efficacy of oral premedication with ivabradine versus propranolol before hypotensive anesthesia with nitroglycerin during endoscopic sinus surgery on reduction of reflex tachycardia.

Secondary aim:

* Compare the safety and incidence of side effects between both drugs.
* Compare the amount of nitroglycerin used, and blood loss between both drugs during endoscopic sinus surgery.

Patients and methods This study will be conducted in the Department of Anesthesia, ENT operating theater, Alexandria University Hospitals after being approved by the Departmental Research and Ethical Committee, and after obtaining informed consents from all patients.

50 Patients, aged from 18 to 39 years, ASA physical status I and II, undergoing endoscopic sinus surgery will be enrolled in the study.

Exclusion Criteria:

* Patients with cardiovascular disease (hypertension, congestive heart failure, and coronary artery disease).
* Patients on beta-blockers.
* Patients with the base line heart rate<60 beats per minute.
* Patients with diabetes mellitus (DM).
* Cerebrovascular insufficiency.
* Coagulation defects.
* History of renal or hepatic insufficiency.
* Hypersensitivity to the study drugs.
* Patients with history of bronchial asthma

The patients will be randomly allocated by simple randomization using a computer programme into two groups by closed envelope technique (having 25 patients in each group):

GROUP (P): will receive oral propranolol (INDERAL® -propranolol hydrochloride Ph. Eur. 10mg manufactured by AstraZeneca Egypt under license of AstraZeneca UK), 10 mg one tablet at 8:00 pm in the evening before the day of the surgery and one 10 mg tablet one hour before the induction of anesthesia.

GROUP (I): will receive oral ivabradine (Procoralan® 5mg manufactured by Servier laboratories, France), 5 mg one tablet at 8:00 pm in the evening before the day of the surgery and one 5 mg tablet one hour before the induction of anesthesia.

Preoperative screening of all patients will include:

1. Demographic data (age, sex).
2. Detailed medical history.
3. Complete physical examination.
4. Routine laboratory investigations:

   * Complete blood picture.
   * Bleeding time and coagulation time.
   * Prothrombin time and activated partial thromboplastin time.
   * Liver enzymes: alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
   * Serum bilirubin (total and direct).
   * Blood urea and serum creatinine.
   * Fasting blood sugar.
5. Chest X-ray.
6. Standard 12 leads electrocardiogram.

Anesthesia:

• All patients will receive the same anesthetic technique.

* Premedication will be standardized for all patients and consists of oral diazepam 5 mg the night before surgery.
* On arrival to operating room, intravenous line will be cited and lactated ringer solution will be infused 4-6 ml/kg/h.
* Before induction of general anesthesia (GA), all patients will be monitored with:
* None-invasive blood pressure (NIBP).
* Electrocardiograph (ECG).
* Pulse oximeter (SpO2).
* After induction of GA, all patients will be monitored with:
* Capnography for end-tidal CO2 (ETCO2).
* Radial artery cannula (G20) for intra-arterial blood pressure monitoring after performing Allen's test.
* Peripheral nerve stimulator (PNS) will be applied on the ulnar nerve for neuromuscular blockade.

Induction and maintenance of anesthesia:

* Anesthesia Will be induced with propofol 2mg/kg iv, fentanyl 1 μg/kg iv and cisatracurium besylate 0.15 mg/kg iv, when TOF count showed disappearance of T1 (0/4) endotracheal intubation with appropriate size will be accomplished and lungs will be mechanically ventilated to maintain the ETCO2 30-35 mmHg.
* Anesthesia will be maintained with inspired isoflurane 1.5 % and cisatracurium besylate top up doses 0.03 mg/kg/30 min will be given guided with TOF count aiming to keep it as 1/4. Airway will be secured by oro-pharyngeal packing and patients will be positioned supine with head up 30°. Dexamethasone 0.2 mg/kg and metoclopramide 10 mg slowly iv will be given as emesis prophylaxis.
* Deliberate hypotension will be induced until completion of the main surgical procedures to achieve a MAP within the target range of 55-65 mm Hg (approximately 30% below a patient's usual MAP), nitroglycerin (1mg/ml) with a dose range 5-20 mcg/min will be added if needed.
* All patients will be operated upon by the same surgical team.
* Bleeding in the surgical field and the quality of the visibility will be assessed subjectively by the surgeon who will be blinded to the infused drug using 6 points scale adapted by Boezaart et al.(25):
* 0= no bleeding.
* 1= slight bleeding so blood evacuation not necessary.
* 2= slight bleeding so sometimes blood has to be evacuated.
* 3= low bleeding so blood has to be often evacuated and operative field is visible for some seconds after evacuation.
* 4= average bleeding so blood has to be often evacuated, and operative field is visible only right after evacuation.
* 5= high bleeding so constant blood evacuation is needed, sometimes bleeding exceeds evacuation and surgery is hardly possible.

The 1st assessment will be 30 min after the beginning of surgery and then every 30 min till the end of surgery.

* As an objective method, the volume of fluid aspirated from the surgical field during surgery will be also measured.
* When blood loss exceed 300 mL, 6% hydroxyethyl starch solutions (Voluven, Fresinius Kabi, Bad Homberg, Germany) will be administered at a 1:1 ratio, and if hematocrit is <27%, a transfusion will be initiated .
* Hypotension (MAP<55 mm Hg) will be treated with ephedrine 15 mg intravenous.
* Bradycardia (HR˂ 50) will be recorded and managed with atropine 0.02mg/kg.
* With termination of surgery, isoflurane will be discontinued, the oropharyngeal pack will be removed and the oropharynx will be suctioned under direct vision using the rigid laryngoscope. The residual cisatracurium will be reversed with neostigmine 0.05 mg/kg iv and atropine 0.02 mg/kg iv when the TOF count is 2/4, trachea will be extubated once the patients showed eye opening and purposeful movement and then patients will be transferred to PACU where BP, SpO2 and ECG will be monitored. O2 supplementation will be provided via face mask.

Measurements:

The following parameters will be measured and will be statistically analyzed between the two studied groups:

1. Demographic data (age and sex).
2. Hemodynamic variables:

   * Mean arterial blood pressure (MABP) in mmHg by invasive monitoring using GE monitor .
   * Heart rate: (beats / minute) using GE monitor.

   Time Points for Hemodynamic Parameter Measurements:
   * Baseline before induction of anesthesia.
   * Before starting the infusion of NTG (baseline)
   * 5 minutes after initiation of NTG
   * Every 30 min throughout deliberate hypotension till termination of NTG infusion.
   * 5 minutes after the end of deliberate hypotension
   * Immediately after extubation in the operating room
   * 60 min after extubation in the PACU
3. The amount of nitroglycerin used:

   * Duration of DH (min(
   * NTG amounts during DH (μg/kg/min).
4. Blood loss and need for blood transfusion:

   * Intraoperative bleeding (mL).
   * Intraoperative autologous blood transfusion (units of packed RBCs).
5. Total urine output (mL).
6. Laboratory investigations:

   * Random blood sugar (RBS)
   * Serum lactate level. Both will be measured immediately after induction of anesthesia, and after discontinuation of deliberate hypotension (NTG infusion).
7. Duration of surgery (the time from start of surgical intervention till its end) (min.).
8. Patients administered ephedrine during DH (n).
9. Events of bradycardia (frequency).
10. Complications need intervention such as bronchospasm, laryngospasm, or vomiting will be recorded and managed.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II, undergoing endoscopic sinus surgery

Exclusion Criteria:

* Patients with cardiovascular disease (hypertension, congestive heart failure, and coronary artery disease).
* Patients on beta-blockers.
* Patients with the base line heart rate<60 beats per minute.
* Patients with diabetes mellitus (DM).
* Cerebrovascular insufficiency.
* Coagulation defects.
* History of renal or hepatic insufficiency.
* Hypersensitivity to the study drugs.
* Patients with history of bronchial asthma

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic changes : | Baseline before induction of anesthesia. - Every 30 min throughout deliberate hypotension till termination of NTG infusion. - 5 minutes after the end of deliberate hypote
  Mean arterial blood pressure (MABP) in mmHg by invasive monitoring using GE monitor .
  • Heart rate: (beats / minute
amount of Blood loss | the procedure time
  Intraoperative bleeding

SECONDARY OUTCOMES:
incidence of Complications | the procedure time
  Complications

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt